CLINICAL TRIAL: NCT03257046
Title: A Randomized, Placebo-Controlled, Double-Blind Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of ITI-214 in Patients With Idiopathic Parkinson's Disease
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ITI-214 in Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-214-105
Record Dates: First submitted 2017-08-14; First posted 2017-08-22 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — ITI-214

STUDY DESIGN:
Intervention Model Description: Multiple rising dose in sequential cohorts of 8 patients randomized in a 6:2 ratio to receive ITI-214 or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 1 mg ITI-214 (Experimental): Administered once daily for 7 days
  Interventions: Drug: ITI-214
- 3 mg ITI-214 (Experimental): Administered once daily for 7 days
  Interventions: Drug: ITI-214
- 10 mg ITI-214 (Experimental): Administered once daily for 7 days
  Interventions: Drug: ITI-214
- 30 mg ITI-214 (Experimental): Administered once daily for 7 days
  Interventions: Drug: ITI-214
- 90 mg ITI-214 (Experimental): Administered once daily for 7 days
  Interventions: Drug: ITI-214
- Placebo (Placebo Comparator): Administered once daily for 7 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ITI-214 — Oral
  Arms: 1 mg ITI-214; 10 mg ITI-214; 3 mg ITI-214; 30 mg ITI-214; 90 mg ITI-214
Other: Placebo — Oral
  Arms: Placebo

SUMMARY:
This is a Phase I/II randomized, double-blind, placebo-controlled, multiple rising dose study in patients with stable idiopathic Parkinson's disease (PD) to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of ITI-214.

ELIGIBILITY:
Major Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease (PD)
* Severity of PD assessed by Hoehn and Yahr Staging score of 1 to 3
* Maintenance on stable PD therapy

Major Exclusion Criteria:

* Clinical signs of dementia
* Suicidal ideation or behavior
* Considered medically inappropriate for study participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with reported or observed treatment-related adverse events | 7 days
  Safety and tolerability

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 7 days
  Pharmacokinetics
Area of the Curve (AUC) | 7 days
  Pharmacokinetics
Motor and non-motor symptoms as assessed by the MDS-UPDRS | 7 days
  Pharmacodynamics

OTHER OUTCOMES:
Exploratory biomarkers | 7 days
  Pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Vanover, PhD, Study Director — Intra-Cellular Therapies, Inc.
Locations (2):
- United States (2):
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Duke Early Phase Research Unit, Durham, North Carolina